CLINICAL TRIAL: NCT02127814
Title: Efficacy and Safety of the Probiotic Lactobacillus Reuteri in the Prevention of Antibiotic Associated-diarrhea and Clostridium Difficile Related Infections in Hospitalized Adult Patients
Brief Title: Lactobacillus Reuteri in the Prevention of Antibiotic Associated-diarrhea and Clostridium Difficile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Alison Steiber, Adjunct profession, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RES504803
Record Dates: First submitted 2010-06-23; First posted 2014-05-01 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Antibiotic-associated Diarrhea; Clostridium Difficile
Keywords: induced diarrhea; Clostridium difficile toxicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri (Experimental)
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Identical Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — One chewable tablet of 1E8 CFU L. reuteri, once per day
  Other Names: BioGaia, Probiotic Chewable Tablets

SUMMARY:
The purpose of this study is to find whether Lactobacillus reuteri prevents antibiotic-associated diarrhea and related Clostridium difficile infections. Subjects will be admitted from the University Hospitals Case Medical Center. They will be randomly assigned to an intervention group receiving L. reuteri or a placebo. Supplementation will occur during antibiotic treatment and for an additional 7 days after cessation of treatment. Data collection will occur at baseline, end of antibiotic use, 7 days after antibiotic cessation, and 21 days after antibiotic cessation. Primary data includes diarrhea instances. Secondary data includes severity of diarrhea, presence of C. difficile toxins, and presence of other GI symptoms.

DETAILED DESCRIPTION:
The data being measured for this study include:

Primary outcome = incidence of diarrhea during and after treatment with antibiotics. An episode of diarrhea is defined as the discrete period between the time when stool output meets or exceeds three soft and unformed or watery bowel movements to the time when formed stools return, which must be at least 48 hours later.

Secondary variables:

1. severity of diarrhea measured as the discrete period between the time when stool output meets or exceeds 3 soft and unformed or watery bowel movements to the time when formed stools return.
2. frequency of stool samples positive for C. Difficile toxin A or B at baseline, when presenting with diarrhea during the study period, and at the follow-up 21 days post-antibiotic-treatment to detect possible clearance of C. Difficile, in patients ingesting L. reuteri versus placebo.
3. frequencies of other gastrointestinal symptoms at 1, 2, and 4 weeks, in the L. reuteri group versus placebo and assessed by the validated Gastrointestinal Symptom Rating Score.

ELIGIBILITY:
Inclusion Criteria:

* Receiving antibiotics for not more than 48 hours prior to enrollment and free from diarrhea
* able to understand and sign informed consent and HIPPA
* available throughout the study period
* subjects should have the mental ability to understand and willingness to fulfill all the details of the protocol

Exclusion Criteria:

* three or more soft and unformed or watery stools per day at admission
* receiving chemotherapy or radiation therapy
* diagnosis of inflammatory bowel disease
* NPO without PO meds
* neutropenia (an absolute neutrophil count (ANC) of less than 1500/microL)
* HIV positive with a CD4+ T-lymphocyte count <400 per mcL blood
* requiring care in an intensive care unit
* status-post bowel resection during hospitalization
* patient's receiving antibiotics four weeks prior to hospitalization
* patient with severe life threatening illness or immunocompromised
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
diarrhea | 28+ days
  Instances of diarrhea

SECONDARY OUTCOMES:
Severity of diarrhea | 28+ days
  measured as the discrete period between the time when stool output meets or exceeds three soft and unformed or watery bowel movements to the time when formed stools return.
Frequency of stool samples positive for C. difficile toxin A and B | baseline, when presenting with diarrhea during the study period, and at the follow-up 21 days
  Frequency of stool samples positive for C. difficile toxin A and B at baseline, when presenting with diarrhea during the study period, and at the follow-up 21 days post antibiotic-treatment to detect possible clearance of C. difficile, in patients ingesting L. reuteri versus placebo.
Frequencies of other gastrointestinal symptoms | 1, 2 and 4 weeks
  Frequencies of other gastrointestinal symptoms at 1, 2 and 4 weeks, in the L. reuteri group versus placebo and assessed by the validated GSRS score (Gastrointestinal Symptom Rating Score).

CONTACTS AND LOCATIONS:
Overall Officials: Alison L Steiber, PhD, RD, LD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States